CLINICAL TRIAL: NCT01385033
Title: A Clinical Trial to Characterize the Performance of [18F]MK-3328 in Subjects With Alzheimer's Disease or Mild Cognitive Impairment, and Healthy Young, and Healthy Elderly Subjects
Brief Title: [18F]MK-3328 as a Possible Novel Positron Emission Tomography (PET) Tracer for the Detection of Brain Amyloid Plaques (MK-3328-002)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 3328-002
Record Dates: First submitted 2011-06-08; First posted 2011-06-29 (Estimated); Results first posted 2014-02-20 (Estimated); Last update posted 2018-11-08 (Actual); Status verified 2018-10

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part I, Healthy Elderly (HE) and AD Participants (Experimental): HE and AD participants will receive a single intravenous (IV) dose of ~150 megabecquerel (MBq) [18F]MK-3328 in Part I of the study
  Interventions: Drug: [18F]MK-3328
- Part II, Healthy Young, HE and AD Participants (Experimental): Healthy Young, HE and AD participants will receive a single IV dose of ~150 megabecquerel (MBq) [18F]MK-3328 in Part II of the study
  Interventions: Drug: [18F]MK-3328
- Part III, Participants with aMCI (Experimental): Participants with aMCI will receive a single IV dose of ~150 megabecquerel (MBq) [18F]MK-3328 in Part III of the study
  Interventions: Drug: [18F]MK-3328

INTERVENTIONS:
Drug: [18F]MK-3328 — IV dose of ~150 megabecquerel (MBq) [18F]MK-3328

SUMMARY:
The purpose of this study is to evaluate radiolabeled [18F]MK-3328 as a PET tracer for estimating the regional distribution and extent of amyloid plaques in participants suffering from amnestic mild cognitive impairment (aMCI) and Alzheimer's Disease (AD) versus healthy young and elderly participants. The study hypotheses will test whether [18F]MK-3328 can discriminate between AD participants and cognitively normal elderly control participants as measured by brain regional tracer uptake.

ELIGIBILITY:
Inclusion Criteria:

All participants:

* Body Mass Index (BMI) between 18 and 35, inclusive, at the pre-screening visit
* Electrocardiogram (ECG) measurements must be clinically acceptable
* Must consent to apolipoprotein E4 (ApoE4) genotyping

Healthy young (HY) and healthy elderly (HE) participants:

* Male or female between the ages of 18 and 45 years (HY) and 65 to 85 years (HE) at pre-screening visit
* Judged to be in good health
* Considered generally cognitively normal

Participants with aMCI or AD:

* Male or female between the ages of 50 and 85 years (aMCI) and 65 to 85 years (AD) at pre-screening visit
* Is in stable medical condition, with existing medical conditions stable for 3 months prior to the pre-screening visit
* Free of any clinically significant disease that would interfere with the study and radiographic evaluations
* Specific cognitive testing requirements for participants aMCI: a history of subjective memory decline with gradual onset and slow progression ≥1 year before Screening, corroborated by an informant; objective impairment in verbal memory as defined by >1 SD below the age adjusted mean for items remembered on the Delayed Word Recall Task of the Alzheimer's Disease Assessment Scale (ADAS) Cog12 at Screening; a global Clinical Dementia Rating (CDR) score of 0.5 and a memory box score of 0.5 or greater at Screening; and an Mini Mental Status Examination (MMSE) score ≥ 24 at Pre-Screening
* Specific cognitive testing requirements for participants with mild-to-moderate AD: MMSE score between 16 and 23, inclusive, at Pre-Screening; modified Hachinski score ≤4 at Screening; meets National Institute of Neurological and Communicative Diseases and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria for probable AD at Screening; Clinical Dementia Rating (CDR) Scale = 0.5, 1 or 2 at Screening; screening magnetic resonance imaging (MRI) scan consistent with a diagnosis of AD
* Participants with AD must have reliable informant/caregiver who is able to accompany the participant to all clinic visits, is able to provide information to study investigator/staff via telephone contact, and agrees to return for per-protocol follow-up visits and procedures
* Participant or participant's legal representative (for participants with AD if the investigator determines that the participant is unable to provide his/her own informed consent) understands the study procedures, and gives written informed consent. For AD participants, the participant's caregiver must also give written informed consent
* Agrees not to participate in any other investigational study that precludes participating in this study

Exclusion Criteria:

* Mentally or legally incapacitated, significant emotional problems at the time of pre-screening visit or expected during the conduct of the study, or has a history of a clinically significant psychiatric disorder over the last 2 years
* Medical history of psychiatric or personality disorders that in the opinion of the investigator and sponsor, affects the ability to participate in the trial
* Has received anti-amyloid agents (e.g., tarenflurbil, tramiprosate) in the 3 months period before screening and has received anti-amyloid antibodies (e.g., bapineuzumab) or anti-amyloid vaccine
* Has participated in MK-3328 PN001 trial
* Has a history of any illness that, in the opinion of the study investigator, might confound the results of the study or poses an additional risk by their participation in the study
* Has had any surgical or medical condition that might significantly alter the distribution, metabolism, or excretion of [18F]-PET tracer
* Has incidental findings on an MRI scan that is pathognomonic for an active disease or pathological process that requires medical intervention
* Has a history of significant infection within 4 weeks prior to study drug administration that in the opinion of the investigator, affects the ability to participate in the trial
* Has an estimated creatinine clearance of ≤30 mL/min based on the Cockcroft-Gault equation
* Has a history of stroke, chronic seizures, or major neurological disorder
* Has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or other diseases that in the opinion of the investigator would prevent them from safely participating in the study
* Has a history of neoplastic disease, except: adequately treated non-melanomatous skin carcinoma or carcinoma in situ of the cervix; other malignancies that have been successfully treated prior to the Pre-Screening visit and appropriate follow-up has revealed no evidence of recurrence; or are highly unlikely to sustain a recurrence for the duration of the study
* Is pregnant, intending to become pregnant within 3 months of ending the study, or is nursing
* Consumes excessive amounts of alcohol, or coffee, tea, cola, or other caffeinated beverages
* Has had major surgery, donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the pre-screening visit
* Has a history of significant multiple and/or severe allergies (including latex allergy), or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food
* Is currently a regular user of any illicit drugs or has a positive screen for drugs with high potential for abuse during the screening period or has a history of drug (including alcohol) abuse within approximately 2 years
* Has a contraindication to undergo PET or MRI including but not limited to claustrophobia, excessive weight or girth, presence of a pacemaker, aneurysm clips, artificial heart valve, ear implant, or metal fragments/foreign objects in the eyes, skin or body
* Has been exposed to ionizing radiation >10 millisievert (mSv) in other research studies within the last 12 months
* Has any disease or condition, or takes any medication that could: interfere with the assessments of safety, tolerability, or biokinetics of the tracer; pose unnecessary risk to the participant; or cause undue discomfort

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-08-19 (Actual); Primary Completion 2012-05-15 (Actual); Study Completion 2012-05-15 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=3328-002&kw=3328-002&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Part II and III were not conducted due to early termination of the study
Groups:
- Alzheimer's Disease (AD) Participants (Part I): AD participants received a single intravenous (IV) dose of ~150 megabecquerel (MBq) [18F]MK-3328, followed by positron emission tomography (PET) imaging of the brain (Part I)
- Healthy Elderly (HE) Participants (Part I): HE participants received a single IV dose of ~150 MBq [18F]MK-3328, followed by PET imaging of the brain (Part I)
- AD Participants (Part II): AD participants received a single intravenous (IV) dose of ~150 megabecquerel (MBq) [18F]MK-3328, followed by PET imaging of the brain (Part II)
- HE Participants (Part II): HE participants received a single IV dose of ~150 MBq [18F]MK-3328, followed by PET imaging of the brain (Part II)
- Healthy Young (HY) Participants (Part II): HY participants received a single IV dose of ~150 MBq [18F]MK-3328, followed by PET imaging of the brain (Part II)
- Amnestic Mild Cognitive Impairment Participants (Part III): Participants with amnestic Mild Cognitive Impairment received a single IV dose of ~150 MBq [18F]MK-3328, followed by PET imaging of the brain (Part III)
Period: Part I
Arm/Group | Alzheimer's Disease (AD) Participants (Part I) | Healthy Elderly (HE) Participants (Part I) | AD Participants (Part II) | HE Participants (Part II) | Healthy Young (HY) Participants (Part II) | Amnestic Mild Cognitive Impairment Participants (Part III)
Started | 6 (These subjects did not participate in Part II or III) | 14 (These subjects did not participate in Part II or III) | 0 | 0 | 0 | 0
Completed | 6 | 14 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part II
Arm/Group | Alzheimer's Disease (AD) Participants (Part I) | Healthy Elderly (HE) Participants (Part I) | AD Participants (Part II) | HE Participants (Part II) | Healthy Young (HY) Participants (Part II) | Amnestic Mild Cognitive Impairment Participants (Part III)
Started | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part III
Arm/Group | Alzheimer's Disease (AD) Participants (Part I) | Healthy Elderly (HE) Participants (Part I) | AD Participants (Part II) | HE Participants (Part II) | Healthy Young (HY) Participants (Part II) | Amnestic Mild Cognitive Impairment Participants (Part III)
Started | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- AD Participants: AD participants received a single IV dose of ~150 MBq [18F]MK-3328, followed by PET imaging of the brain
- HE Participants: HE participants received a single IV dose of ~150 MBq [18F]MK-3328, followed by PET imaging of the brain
- Total: Total of all reporting groups
Arm/Group | AD Participants | HE Participants | Total
Number analyzed (Participants) | 6 | 14 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (5.8) | 71.9 (5.8) | 69.5 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 10
  Male | 3 | 7 | 10

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Receiver Operating Curve (AUC of ROC) for Distinguishing Between AD and HE Participants Based on Brain Cortical [18F]MK-3328 Standard Uptake Value Ratio (SUVR)
Description: Using PET brain images acquired after dosing, regions of interest (ROIs) are drawn in identified brain areas. The ROIs are projected onto all frames of the dynamic PET scans in order to generate [18F]MK-3328 tissue time-activity curves (TACs). SUVR is calculated as the ratio of the average [18F]MK-3328 uptake over 60-90 minutes post dose in the target brain region and the cerebellum. Cortical SUVR is determined, which is a mean SUVR derived from SUVR from multiple brain regions (frontal cortex, parietal cortex, anterior cingulate gyrus, posterior cingulate gyrus, temporal cortex, lateral temporal cortex and occipital cortices). The receiver operating curve (ROC) for determining whether a participant is in HE or AD group by using cortical SUVR values is determined. The ROC is a plot of sensitivity on the y-axis versus 1-specificity (false positive rate) on the x-axis for the range of cortical SUVR threshold values. The AUC of ROC is determined.
Time Frame: 60-90 minutes post dose
Population: The study was terminated early before completion of Part I. Given the low number of enrolled AD participants (6 of up to 15 planned in Part I), the interim analysis for futility in Part I was not conducted and the potential of [18F]MK-3328 to distinguish between AD and HE participants was not assessed.
Groups:
- AD and HE Participants: AD and HE participants received a single IV dose of ~150 MBq [18F]MK-3328, followed by PET imaging of the brain
Arm/Group | AD and HE Participants
Number analyzed (Participants) | 0

2. Primary Outcome: Brain Cortical [18F]MK-3328 SUVR in AD Participants and HE Participants
Description: Using PET brain images acquired after dosing, ROIs are drawn in identified brain areas. The ROIs are projected onto all frames of the dynamic PET scans in order to generate [18F]MK-3328 tissue TACs. SUVR is calculated as the ratio of the average [18F]MK-3328 uptake over 60-90 minutes post dose in the target brain region and the cerebellum. Cortical SUVR is reported, which is a mean SUVR derived from SUVR from multiple brain regions (frontal cortex, parietal cortex, anterior cingulated gyrus, posterior cingulated gyrus, temporal cortex, lateral temporal cortex and occipital cortices). A trimming procedure will be applied to remove the sub-population of HE participants who have positive amyloid plaque burden. The 1st and 2nd quartiles of the cortical SUVR distribution, Q1 and Q2, are computed for HE data; values with SUVR ≥(Q2-Q1)*3 are removed before calculation of HE mean (trimmed) and standard deviation (SD)(trimmed).
Time Frame: 60-90 minutes post dose
Population: The study was terminated early before completion of Part I. Given the low number of enrolled AD participants (6 of up to 15 planned in Part I), the interim analysis for futility in Part I was not conducted and the determination of brain cortical [18F]MK-3328 SUVR values in AD and HE participants was not performed.
Arm/Group | AD Participants | HE Participants
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Amyloid Plaque Burden Threshold Determined by the Trimmed HE Sample Mean and SD Brain Cortical [18F]MK-3328 SUVR
Description: Using PET brain images acquired after dosing, ROIs are drawn in identified brain areas. ROIs are projected onto all frames of the dynamic PET scans in order to generate [18F]MK-3328 tissue TACs. SUVR is calculated as the ratio of the average [18F]MK-3328 uptake over 60-90 minutes post dose in the target brain region and the cerebellum. Cortical SUVR is determined, which is a mean SUVR derived from SUVR from multiple brain regions. The 1st and 2nd quartiles of the cortical SUVR distribution, Q1 and Q2, are computed for HE data; values with SUVR ≥(Q2-Q1)*3 are removed before calculation of HE mean (trimmed) and SD (trimmed). This step is performed to remove HE participants with positive plaque burden. Using HE data, the threshold for classification of plaque burden as positive/negative will be calculated as mean (trimmed) + k*SD (trimmed). Value of k will be chosen to fine tune sensitivity/specificity, with specificity of at least 0.9 in the sub-group remaining after trimming of data.
Time Frame: 60-90 minutes post dose
Population: The study was terminated early before completion of Part I. Given the low number of enrolled AD participants (6 of up to 15 planned in Part I), the interim analysis for futility in Part I was not conducted and the determination of an amyloid plaque burden threshold using PET imaging data obtained after [18F]MK-3328 administration was not performed.
Arm/Group | HE Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 14 days after last dose
Groups:
- All Study Participants: Participants received a single IV dose of ~150 MBq [18F]MK-3328, followed by PET imaging of the brain
Arm/Group | All Study Participants
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 4/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Study Participants (N=20)
Diarrhoea (Gastrointestinal disorders) | 1
Injection site pain (General disorders) | 1
Sinusitis (Infections and infestations) | 1
Presyncope (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication timelines.